CLINICAL TRIAL: NCT00011115
Title: Weight Loss Motivations and Long-term Weight Loss
Brief Title: Motivations for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Model: Factorial | Purpose: Treatment
Other Study IDs: Klem-Motivation (completed); R01DK058387 (NIH)
Record Dates: First submitted 2001-02-09; First posted 2001-02-09 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: overweight
MeSH Terms: conditions — Obesity; Overweight

INTERVENTIONS:
Behavioral: Weight loss motivations

SUMMARY:
This study tests the effects of emphasizing different motivations for wanting to lose weight on weight loss maintenance in women. At the start of the study, participants will be weighed and will complete questionnaires about their health, weight history, eating and exercise habits, body satisfaction and mood. Participants will then be randomly assigned to 1 of 4 treatments. Participants in all 4 groups will receive information on topics related to eating and exercise, and will receive calorie and fat intake goals, and exercise goals. The 4 treatments will differ in the emphasis given to various reasons for wanting to lose weight. At 6, 12 and 18 months after enrollment, participants will again have weights measured and fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index greater than or equal to 27 and less than or equal to 35
* Rating both physical appearance and health concerns as important motivations for weight loss
* Successful completion of a food and exercise diary over a 5-day period

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2001-09; Study Completion 2003-05

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh School of Medicine, Dept of Psychiatry, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kalarchian MA, Levine MD, Klem ML, Burke LE, Soulakova JN, Marcus MD. Impact of addressing reasons for weight loss on behavioral weight-control outcome. Am J Prev Med. 2011 Jan;40(1):18-24. doi: 10.1016/j.amepre.2010.09.019. PMID 21146763